CLINICAL TRIAL: NCT03518580
Title: Using Ecological Momentary Assessment to Examine Within-person Variations in Daily Experiences of Active Life Engagement in Relation to Health-related Outcomes Among Community-dwelling Chinese Older Adults
Brief Title: Active Life Engagement in Relation to Health-related Outcomes Among Community-dwelling Chinese Older Adults
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Vivian W.Q. Lou, Associate Professor, The University of Hong Kong
Other Study IDs: EA1706016
Record Dates: First submitted 2018-03-22; First posted 2018-05-08 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Aging
Keywords: mobile technology; real-time assessment; active life engagement

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: real-time assessment of biopsychosocial functioning — the participants were asked to provide biopsychosocial data using the mobile device

SUMMARY:
This study aims to examine within-person variations of different contexts (time, physical, psychosocial and affective) of active life engagement, and how these variations predict a set of physiological indicators and health-related outcomes among community-dwelling older people. Specifically, this study has the following objectives.

Objective 1: To investigate within-person variations in different contexts (i.e., time, physical, psychosocial, and affective) of active life engagement and interactions of these contexts.

Objective 2: To examine how within-person variations in different contexts (i.e., time, physical, psychosocial, and affective) of active life engagement and interactions of these contexts may associate with a set of cardiovascular indicators measured on daily basis.

Objective 3: To examine how within-person variations in different contexts (i.e., time, physical, psychosocial, and affective) of active life engagement and interactions of these contexts may associate with a set of health-related outcomes (e.g., physical functioning, depression, health-related quality of life).

DETAILED DESCRIPTION:
1. Participants

This study will recruit 70 participants from the community with the help from staffs from community service center. Investigators recruited participants who aged 60 or older and lived in the community independently, and screened participants for eligibility based on the following exclusionary criteria: (1) unable to complete brief survey presented in mobile devices (e.g., have severe visual deficits or other self-report difficulty reading the screen), (2) diagnosed with a cognition disorder, (4) diagnosed with a mental disorder.

Study protocol

I. Self-administered questionnaire survey

All the participants will be asked to complete the baseline self-administrated survey on line (in some cases, participants could be organized to complete the survey under the guide of the research staff).

II. Training sessions/orientation

All the eligible participants will be invited to attend the training session/orientation. The research staff will assign each participant a Android phone installed with a researcher-developed application and a mobile-electrocardiogram (ECG) recording device. The participants will be briefed on its basic functions and how to use the application and device to provide data. The whole session will take steps proactively to increase participants' confidence and comfort with using the electronic band and the real-time assessment application through in-person training and mutual support between participants. Detailed take-home handbook (hardcopy or electronic version) that cover the use guidelines of the electronic bans and the real-time assessment application, and troubleshooting help, will be distributed to participants. Then, two warm-up days prior to the main study will be conducted and on-call help will be provided.

III. Real-time assessment survey of daily experiences

The real-time assessment application will allow each user to register a personal account, and to define their person-specific time-frame for the procedure, in specific, the start and the end time in a typical day they accept the signaling. The time frame will basically cover the user's waking hours (approximately 7 ± 3 hours). Within the defined time frame, the mobile device with the application will randomly prompt the user to complete a report for 6 times. The minimum and the maximum time between two consecutive signals will be 30 and 150 minutes respectively. The device will correctly record each response time once sending the signal. If the device receives no response for over 20 minutes, substitute prompts will be automatically sent every 5 minutes for 2 times. If still no response, a missing will be recorded. This procedure will be repeated on 7 consecutive days, with different random patterns for each day. For answering one signaling report, it will take approximately 3 to 5 minutes for most users (a total of less than 30 min per day). The content of report will be the same each time, which will comprise questions on engagement in daily activities, individual distractions, mood, and social systems.

IV. Physiological data provision

Physiological data will be collected concurrently during the 7 consecutive days for real-time data collection. All participants will be required to carry the mobile-ECG device assigned to them during the whole process of data collection. They will use the smartphone-based application and the mobile-ECG device to provide a 30-second ECG recording for six times each day.

V. In-person follow-up survey

All participants will be asked to complete the open-ended questions focusing on the feasibility/acceptability of the method.

No drug usage and medical treatment will be involved in the study. Intensive assessment do not impose any physical or medical risk to participants. The only possible problem is that the intensive assessment may interfere with the participants' normal daily routines. Participants can voluntarily drop out the study at any time, without giving any reason.

Data analyses:

Intra-individual variability in the activity engagement will be analyzed by calculating the standard-deviation for each participant's timing of each domains of engagement resulting in an intra-individual standard deviation (iSD). In order to model within-person change and between-person factors simultaneously, two alternative statistical methods, namely, time series analysis and random coefficient multilevel modelling will be used. Multiple hierarchical regression analyses will be conducted with activity indicators predicting health and well-being outcomes.

ELIGIBILITY:
Inclusion Criteria:

* aged between 50-70; lived in the community independently; volunteer to participate in this study

Exclusion Criteria:

* unable to complete brief survey presented in mobile devices (e.g., have severe visual deficits or other self-report difficulty reading the screen);
* diagnosed with a cognition disorder or a mental disorder (e.g., major depressive disorder);
* diagnosed with hypertension or history of chronic disease with a cardiovascular component (e.g., diabetes);
* use of cardiovascular prescription medication, consumption of more than 10 alcoholic beverages a week.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy aging population living in the urban areas of a site city, Changsha in the central part of China.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2017-07-02 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-03-05 (Actual)

PRIMARY OUTCOMES:
Momentary positive and negative emotion | one week
  The extent to which the participant feel happy, excited, calm, sad, anxious, irritated, sleepy, alert, quiet, and lonely at the assessment time (0 = not at all to 4 = very much).

CONTACTS AND LOCATIONS:
Overall Officials: Vivian Lou, PhD, Principal Investigator — Sau Po Center on Ageing, HKU
Locations (1):
- Sau Po Center on Ageing HKU, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Data collected in this study will be published and submitted to academic journals to share with other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Between 2018 and 2021, the data will become available.
Access Criteria: Upon request from the academic journals.

REFERENCES:
- [Derived] Fang B, Li D, Chen B, Huang J, Hou Y, Liu H. Perceived Support Protects Against Negative Affective Experiences of Momentary Solitude: An Ecological Momentary Assessment Study. J Gerontol B Psychol Sci Soc Sci. 2022 Dec 29;77(12):2170-2181. doi: 10.1093/geronb/gbac081. PMID 35678188